CLINICAL TRIAL: NCT01860287
Title: The Effects of Buprenorphine on Responses to Verbal Tasks
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UCIRB-130197
Record Dates: First submitted 2013-05-06; First posted 2013-05-22 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-04

CONDITIONS: Basic Science
Keywords: opioid; subjective; stress; buprenorphine
MeSH Terms: interventions — Buprenorphine; Administration, Sublingual

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo group (Placebo Comparator): Healthy volunteers receive placebo during session (within-subjects design).
  Interventions: Drug: Placebo
- buprenorphine (0.2 mg) group (Experimental): Healthy volunteers receive buprenorphine (0.2 mg) during session (within-subjects design).
  Interventions: Drug: Buprenorphine 0.2 MG Sublingual Tablet
- buprenorphine (0.4 mg) group (Experimental): Healthy volunteers receive buprenorphine (0.4 mg) during session (within-subjects design).
  Interventions: Drug: Buprenorphine 0.4 MG Sublingual Tablet

INTERVENTIONS:
Drug: Buprenorphine 0.2 MG Sublingual Tablet — This is a within-subjects, double-blind, placebo-controlled experiment during which each participant will receive sublingual buprenorphine (0.2)
  Arms: buprenorphine (0.2 mg) group
Drug: Placebo — This is a within-subjects, double-blind, placebo-controlled experiment during which each participant will receive a placebo
  Arms: Placebo group
Drug: Buprenorphine 0.4 MG Sublingual Tablet — This is a within-subjects, double-blind, placebo-controlled experiment during which each participant will receive sublingual buprenorphine (0.4)
  Arms: buprenorphine (0.4 mg) group

SUMMARY:
In this study, the investigators will examine the effects of buprenorphine, as compared to placebo, upon physiological, subjective, and hormonal responses to a stressful speech task and a non-stressful control task in healthy adults. There is strong evidence in support of the role of endogenous opioids and opiates in mediating social behavior in humans and other animals, and particularly, in social distress. Recently it has been shown that buprenorphine, a partial mu-opioid agonist, reduces sensitivity to recognition of fearful facial expressions in humans. Here, the investigators propose to further explore the role of the opioid system in mediating stress responses in humans through the use of buprenorphine. The investigators hypothesize that buprenorphine with reduce both physiological and subjective measures of stress.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* ages 18-40 years
* high school education
* fluent in English

Exclusion Criteria:

* history of adverse drug reactions
* taking oral contraceptives or planning to become pregnant
* taking any medications
* smokers
* night shift workers
* drink more than 4 alcoholic or caffeinated drinks per day

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, Ph.D., Principal Investigator — University of Chicago; Jerome Jaffe, M.D., Study Chair — University of Maryland
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: Healthy volunteers receive placebo
- 0.2 Buprenorphine: Healthy volunteers will receive 0.2 mg of buprenorphine
- 0.4 mg Buprenorphine: Healthy volunteers will receive 0.4 mg of buprenorphine
Period: Overall Study
Arm/Group | Placebo Group | 0.2 Buprenorphine | 0.4 mg Buprenorphine
Started | 18 | 15 | 15
Completed | 18 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Buprenorphine (0.2 mg) Group | Buprenorphine (0.4 mg) Group | Total
Number analyzed (Participants) | 18 | 15 | 15 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 15 | 15 | 48
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 4 | 16
  Male | 12 | 9 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: Subjective Effects as Assessed by Score on "Feel Drug", "Feel High", "Like Drug", and "Want More" Subscales of the Drug Effects Questionnaire Subjective Responses to Stress With and Without Buprenorphine
Description: The Drug Effects Questionnaire (DEQ) is a visual analog scale questionnaire that assesses the extent to which subjects experience four subjective states: "Feel Drug", "Feel High", and "Want More". The "Feel Drug", "Feel High", "Like Drug", and "Want More" subscales are reported. All subscales are scored on a visual analogue scale (scroll bar on computer screen) ranging from 0 -100. 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome.
Time Frame: End of study - (Pre-administration of drug or placebo (Time 0), and approx 210 minutes after drug/placebo admin), End of study (210 min) shown
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Group | 0.2 Buprenorphine | 0.4 mg Buprenorphine
Number analyzed (Participants) | 18 | 15 | 15
units on a scale
  Feel Drug | 13.57 (2.1) | 36.57 (4.5) | 59.89 (1.55)
  Like Drug | 9.4 (1.2) | 43.27 (3.6) | 56.25 (4.22)
  Feel High | 6.0 (1.5) | 27.27 (2.5) | 41.69 (3.45)
  Want More | 4.27 (1.3) | 12.47 (1.9) | 21.57 (1.96)

ADVERSE EVENTS:
Time Frame: 6 days for each intervention
Arm/Group | Placebo Group | 0.2 Buprenorphine | 0.4 mg Buprenorphine
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes